



**Title of Project:** "Success and survival of root canal treated tooth restored using ceramic onlays"

Name of Researcher: Noushad Rahim, Rupert Austin, Prof Francesco Mannocci

Name of Statistician: A. Manoharan

Please find below the power calculation statement.

## **Power Calculation Statement:**

The sample size calculation for this study was based on chi-test for testing the association between tooth surface lost (<33%, 33-66% and >66%) and Root Canal Treatment status (Success or Failure). A study with an effect size of 0.3 and a power of 80% will require a total sample of 108 to test the association at 5% levels using two tailed test. The power calculation was carried out using Gpower 3.1.7.

Regards,
A.Manoharan.
<a href="mailto:manoharan.1.andiappan@kcl.ac.uk">manoharan.1.andiappan@kcl.ac.uk</a>
12/04/2017